CLINICAL TRIAL: NCT06436027
Title: Molecular Diagnosis of Heart Allograft Rejection Using Intra-Graft Targeted Gene Expression Profiling.
Acronym: Nano-Heart
Status: Completed | Type: Observational
Sponsor: Paris Translational Research Center for Organ Transplantation (Other)
Collaborators: Cedars Sinai Medical Center, Los Angeles, USA (Unknown); University of Padova (Other)
Responsible Party: Sponsor
Other Study IDs: NANOHEART
Record Dates: First submitted 2024-05-14; First posted 2024-05-30 (Actual); Last update posted 2024-05-30 (Actual); Status verified 2024-05

CONDITIONS: Heart Transplant Rejection
Keywords: molecular biology; allograft rejection; endomyocardial biopsy; pathology; precision diagnosis; heart transplantation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Biospecimen Retention: Samples Without DNA — Use of formalin-fixed paraffin-embedded endomyocardial biopsies collected prospectively as part of the standard clinical care of heart transplant recipients.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Development cohort: Random selection of 80% of the overall cohort.
  Interventions: Diagnostic Test: Nano-Heart tool: Intra-Graft Targeted Gene Expression Profiling
- Validation cohort: Random selection of 20% of the overall cohort.
  Interventions: Diagnostic Test: Nano-Heart tool: Intra-Graft Targeted Gene Expression Profiling

INTERVENTIONS:
Diagnostic Test: Nano-Heart tool: Intra-Graft Targeted Gene Expression Profiling — Targeted molecular profiling will be performed on formalin-fixed paraffin-embedded (FFPE) endomyocardial biopsies using the NanoString nCounter technology. A consortium-approved consensual targeted panel including 770 genes, developed by the Banff Molecular Diagnostics Working Group (MDWG) will be used.

SUMMARY:
The goal of this observational study is to develop and validate a molecular heart rejection diagnostic system based on targeted transcriptome as a novel monitoring companion tool for heart allograft precision diagnostics applicable to formalin-fixed paraffin-embedded endomyocardial biopsies.

The primary outcome will be the biopsy-proven rejection, that will be predicted with molecular classifiers (cellular and antibody-mediated rejection scores).

DETAILED DESCRIPTION:
Heart transplantation (HTx) remains the most valuable therapeutic option for patients with end-stage heart failure refractory to optimal medical therapy. Despite major improvements in immunosuppression and transplant care, acute and chronic rejection-induced allograft injuries remain one of the leading causes of mortality and morbidity after heart transplantation, thus limiting recipients' life expectancy. An improvement in the overall management of rejection remains an unmet medical need. As a first step, a precise diagnosis of rejection is crucial to guide patient care and optimize management.

Nowadays, the diagnosis of cardiac rejection relies exclusively on the pathological assessment of endomyocardial biopsies (EMBs) by identifying and grading cellular infiltrates and myocardial damage. While important advances have been made in the standardization of the rejection diagnosis, pathology remains an imperfect gold-standard, particularly due to the inter-observer variability, sample bias and the use of qualitative or semi-quantitative scales that oversimplify complex phenotypes. Additionally, disease severity, degree of myocardial injury and progression stage are crucial pieces of information poorly captured by the current working formulations. All these limits represent major barriers to achieve a precise and reliable diagnosis of rejection.

In this context, gene expression profiling analysis of fresh myocardial samples retrieved during an extra-core biopsy and using a whole transcriptome approach arose as a potential objective companion tool of pathology to refine the diagnosis of rejection. However, important drawbacks have limited the routine clinical applicability of whole-transcriptome based molecular diagnosis including extra-core sampling bias, low reproducibility, technical and analytical heaviness, with costs and sample turn-around that is not compatible with a clinical setting.

Recent technologies may overcome this limitation by allowing analysis of the same tissue used for histology assessment. Targeted molecular profiling applicable to formalin-fixed paraffin-embedded (FFPE) endomyocardial biopsies may allow the implementation of molecular diagnosis into the clinical routine. Recently, we have shown that the Banff Human Organ Transplant Panel (B-HOT) panel, a consortium-approved consensual targeted panel including 770 genes, developed by the Banff Molecular Diagnostics Working Group, accurately captured key molecular patterns of antibody-mediated rejection (AMR) in heart allograft biopsies and may serve as a proxy to whole transcriptome-based analysis.

The aim of the present study is therefore to identify gene expression signatures for AMR and acute cellular rejection in heart transplantation and to develop and validate a molecular heart rejection diagnostic system based on targeted transcriptome as a novel monitoring companion tool for heart allograft precision diagnostics applicable to FFPE-EMB.

ELIGIBILITY:
Inclusion Criteria:

* heart transplant recipients ≥ 18 years old
* at least one endomyocardial biopsy performed as part of routine clinical care
* biopsy performed at least ≥ 1 month post transplant and less that 10-year post-transplant
* written informed consent

Exclusion Criteria:

* age below 18 years old

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: We designed an international multicenter study, building a deep phenotyped cohort of heart transplant recipients recruited at 4 referral centers (Pitié-Salpêtrière and Georges Pompidou hospitals in Paris, Center Gallucci of the University General Hospital of Padova and the Cedars Sinai Medical Center in Los Angeles, USA).
Sampling Method: Probability Sample
Enrollment: 496 (Actual)
Dates: Start 2021-11-10 (Actual); Primary Completion 2023-12-15 (Actual); Study Completion 2023-12-15 (Actual)

PRIMARY OUTCOMES:
Biopsy-proven rejection: acute cellular-rejection and antibody-mediated rejection. | 1 month
  Prediction performances of the molecular classifiers (cellular and antibody-mediated rejection scores) to predict biopsy-proven rejection: diagnostic accuracy, Receiver Operating Characteristic - area under the curve, Precision Recall - area under the curve, Brier score, F1 score.

SECONDARY OUTCOMES:
Discrepancies between molecular and pathology diagnosis of rejection. | 1-month
  Confusion matrix, detailed review of the cases.

CONTACTS AND LOCATIONS:
Overall Officials: Alexandre Loupy, MD, PhD, Study Director — Paris Translational Research Center for Organ Transplantation; Guillaume Coutance, MD, PhD, Principal Investigator — Paris Translational Research Center for Organ Transplantation
Locations (3):
- Cedars Sinai Medical Center, Los Angeles, California, United States
- Paris Translational Research Center for Organ Transplantation, Paris, France
- Center Gallucci of the University General Hospital of Padova, Padua, Italy

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Berry GJ, Burke MM, Andersen C, Bruneval P, Fedrigo M, Fishbein MC, Goddard M, Hammond EH, Leone O, Marboe C, Miller D, Neil D, Rassl D, Revelo MP, Rice A, Rene Rodriguez E, Stewart S, Tan CD, Winters GL, West L, Mehra MR, Angelini A. The 2013 International Society for Heart and Lung Transplantation Working Formulation for the standardization of nomenclature in the pathologic diagnosis of antibody-mediated rejection in heart transplantation. J Heart Lung Transplant. 2013 Dec;32(12):1147-62. doi: 10.1016/j.healun.2013.08.011. PMID 24263017
- [Background] Halloran PF, Venner JM, Madill-Thomsen KS, Einecke G, Parkes MD, Hidalgo LG, Famulski KS. Review: The transcripts associated with organ allograft rejection. Am J Transplant. 2018 Apr;18(4):785-795. doi: 10.1111/ajt.14600. Epub 2017 Dec 23. PMID 29178397
- [Background] Halloran PF, Potena L, Van Huyen JD, Bruneval P, Leone O, Kim DH, Jouven X, Reeve J, Loupy A. Building a tissue-based molecular diagnostic system in heart transplant rejection: The heart Molecular Microscope Diagnostic (MMDx) System. J Heart Lung Transplant. 2017 Nov;36(11):1192-1200. doi: 10.1016/j.healun.2017.05.029. Epub 2017 May 29. PMID 28662985
- [Background] Mengel M, Loupy A, Haas M, Roufosse C, Naesens M, Akalin E, Clahsen-van Groningen MC, Dagobert J, Demetris AJ, Duong van Huyen JP, Gueguen J, Issa F, Robin B, Rosales I, Von der Thusen JH, Sanchez-Fueyo A, Smith RN, Wood K, Adam B, Colvin RB. Banff 2019 Meeting Report: Molecular diagnostics in solid organ transplantation-Consensus for the Banff Human Organ Transplant (B-HOT) gene panel and open source multicenter validation. Am J Transplant. 2020 Sep;20(9):2305-2317. doi: 10.1111/ajt.16059. Epub 2020 Jun 27. PMID 32428337
- [Background] Giarraputo A, Coutance G, Aubert O, Fedrigo M, Mezine F, Zielinski D, Mengel M, Bruneval P, Duong van Huyen JP, Angelini A, Loupy A. Banff Human Organ Transplant Consensus Gene Panel for the Detection of Antibody Mediated Rejection in Heart Allograft Biopsies. Transpl Int. 2023 Sep 4;36:11710. doi: 10.3389/ti.2023.11710. eCollection 2023. PMID 37745639
- [Background] Coutance G, Zouhry I, Racape M, Drieux F, Viailly PJ, Rouvier P, Francois A, Chenard MP, Toquet C, Rabant M, Berry GJ, Angelini A, Bruneval P, Duong Van Huyen JP. Correlation Between Microvascular Inflammation in Endomyocardial Biopsies and Rejection Transcripts, Donor-specific Antibodies, and Graft Dysfunction in Antibody-mediated Rejection. Transplantation. 2022 Jul 1;106(7):1455-1464. doi: 10.1097/TP.0000000000004008. Epub 2021 Dec 21. PMID 34954735
- [Background] Duong Van Huyen JP, Fedrigo M, Fishbein GA, Leone O, Neil D, Marboe C, Peyster E, von der Thusen J, Loupy A, Mengel M, Revelo MP, Adam B, Bruneval P, Angelini A, Miller DV, Berry GJ. The XVth Banff Conference on Allograft Pathology the Banff Workshop Heart Report: Improving the diagnostic yield from endomyocardial biopsies and Quilty effect revisited. Am J Transplant. 2020 Dec;20(12):3308-3318. doi: 10.1111/ajt.16083. Epub 2020 Jun 28. PMID 32476272